CLINICAL TRIAL: NCT01655316
Title: Oral Verapamil in Acute Paroxysmal Supra Ventricular Tachycardia(PSVT) Recurrence Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 16062
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Paroxysmal Supraventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Verapamil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Verapamil (Experimental): 40 mg Verapamil Per Oral
  Interventions: Drug: Verapamil

INTERVENTIONS:
Drug: Verapamil

SUMMARY:
PSVT is a common rhythm disorder in emergency department which can be recurrent in some cases.

Intravenous Adenosine is the drug of choice in PSVT control in acute settings but is a very short acting agent.

Providing a complementary medication to decrease the rate of recurrence of PSVT after its initial control will be promising.

This study evaluates the role of the oral Verapamil in recurrence control of PSVT in emergency situations.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old
* PSVT on emergency department presentation

Exclusion Criteria:

* Instability in hemodynamic status
* Allergy to Verapamil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Recurrence Control | 2 hours